CLINICAL TRIAL: NCT06167278
Title: INDIRECT BONDING ACCURACY OF TWO DIFFERENT 3D PRINTED DIGITAL TRANSFER TRAYS: A RANDOMIZED CLINICAL TRIAL
Brief Title: Indirect Bonding Accuracy of 3D Printed Digital Transfer Trays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Marmaraortho1
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Orthodontics; Bracket Bonding; Indirect Bonding; Digital Indirect Bonding Transfer Tray; Accuracy of Bracket Positioning
Keywords: 3D printed indirect bonding transfer tray

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shell tray group (Experimental)
  Interventions: Other: Indirect bonding with two different digital bracket bonding transfer tray
- Bar tray group (Experimental)
  Interventions: Other: Indirect bonding with two different digital bracket bonding transfer tray

INTERVENTIONS:
Other: Indirect bonding with two different digital bracket bonding transfer tray — To achieve more precise and predictable result is the common aim in contemporary treatment. Digital indirect bonding (IDB) is used for this purpose in orthodontic treatment. The aim of this study is to compare the transfer accuracy of two different IDB trays.
  Digital IDB was performed on a total of 30 patients, using one of the two designs: shell and bar trays; with 15 patients in each group. Trays were designed with the Appliance Designer software (3Shape A/S, Copenhagen, Denmark) as shell and bar types.

SUMMARY:
The goal of this study is to compare the bracket transfer accuracy of two frequently used 3D printed indirect bonding trays.

This is an interventional study. Participants have 3-6mm crowding without tooth loss and deformity. It is planned to be 2 groups in the study. Each group will include 15 participants. Indirect bonding will be applied with shell and bar designs that are frequently used. Brackets will be bonded from second premolar to other side's second premolar of upper and lower jaw. Bracket transfer accuracy of two different trays will be compared with planned position and each other.

DETAILED DESCRIPTION:
There are planned to be 2 groups in the study. Each group will include 15 participants. The patients who apply for orthodontic treatment will be included in this study. inclusion criteria: patients between age of 17-30, in complete permanent dentition, have mild to moderate (3-6mm) crowding according to Little's irregularity index, good oral hygiene and periodontal health. The exclusion criteria were patients needing treatment with extraction, having shape anomaly, deficiency, fractures, crowns or abrasions in their teeth. Informed and written consent forms will be obtained from each patient for experimentation.

Intraoral scans with the 3Shape device (3Shape TRIOS, Copenhagen, Denmark) are routinely recorded from the patients whose treatment will begin before treatment. Bracket positions will be adjusted on the scan images using 3Shape OrthoAnalyzer 2015 software. Then, the bracket model will be transferred to the Appliance Designer software program, 2 types of transfer trays will be designed and produced with the 3D printer in the clinic. Patients will be indirectly bracketed with the produced transfer trays and intraoral scan recordings will be taken again after bracketing. This image and the images where the brackets are placed in the software will be overlaid with the GOM Inspect software (GOM GmbH, Braunschweig, Germany) and the deviations will be calculated for both transfer trays and the differences will be compared.

The measurements to be performed are: linear: mesiodistal, buccolingual, incisogingival; angular: torque, angulation, rotation. Measurements will be calculated separately for all teeth.

None of these steps deviate from the routine treatment protocol and none of the procedures are harmful or invasive for the patient.

ELIGIBILITY:
Inclusion Criteria:

Patients between age of 17-30, in complete permanent dentition, have mild to moderate (3-6mm) crowding according to Little's irregularity index, good oral hygiene and periodontal health.

Exclusion Criteria:

Patients needing treatment with extraction, having shape anomaly, deficiency, fractures, crowns or abrasions in their teeth.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of bracket position | 15 days
  Angular (torque, tip, angulation) and linear (mesiodistal, buccolingual, occlusogingival) differences will be compared between the bonded intraoral scans taken immediately after IDB and the virtually bracketed model prepared in the Ortho Analyzer software (3Shape A/S, Copenhagen, Denmark) using the open source GOM inspect software (GOM GmbH, Braunschweig, Germany).

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No